CLINICAL TRIAL: NCT06752239
Title: Prophylactic Radiotherapy Optimization for Enhanced Thyroid Function Protection in Nasopharyngeal Carcinoma (PROTECT-NPC): A Multicenter, Non-Inferiority, Open-Label, Randomized Controlled Phase III Clinical Trial
Brief Title: Prophylactic Radiotherapy Optimization for Enhanced Thyroid Function Protection in NPC
Acronym: PROTECT-NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jingao Li, PI, Jiangxi Provincial Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-NPC
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Nasopharyngeal Carcinoma; Quality of Life; Thyroid Diseases; Radiotherapy Side Effect; Radiotherapy
Keywords: Nasopharyngeal Carcinoma; Quality of Life; Thyroid Function Protection; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Thyroid Diseases; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard delineation (Active Comparator): The medial edge of the level III-IVa lymphatic drainage areas was the medial edge to encompass the common carotid artery. And the anterior boundary of the level III-IVa drainage area as the anterior edge of the common carotid artery or posterior edge of the thyrohyoid muscle rather than the anterior edge of the sternocleidomastoid muscle or the posterior third of the thyrohyoid muscle, to reduce thyroid radiation exposure
  Interventions: Radiation: Standard delineation
- Modified delineation (Experimental): The medial edge of the level III-IVa lymphatic drainage areas was redefined to the lateral edge of the common carotid artery, sparing the common carotid artery area. The anterior boundary of the level III-IVa drainage area as the anterior edge of the common carotid artery or posterior edge of the thyrohyoid muscle, rather than the anterior edge of the sternocleidomastoid muscle or the posterior third of the thyrohyoid muscle, to reduce thyroid radiation exposure.
  Interventions: Radiation: Modified delineation

INTERVENTIONS:
Radiation: Modified delineation — Modified delineation (MD) of cervical lymphatic drainage areas, sparing the common carotid artery within the clinical target volume (CTV)
  Other Names: MD
  Arms: Modified delineation
Radiation: Standard delineation — Standard delineation
  Arms: Standard delineation

SUMMARY:
This study is a multicenter, non-inferiority, open-label, randomized controlled Phase III clinical trial. It aims to compare the efficacy of modified delineation radiotherapy (experimental group) versus standard delineation radiotherapy (control group) in the prophylactic irradiation of neck lymphatic drainage areas III/IVa in nasopharyngeal carcinoma. The study evaluates the incidence of primary hypothyroidism, quality of life, and adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-70 years; 2. Pathologically confirmed nasopharyngeal carcinoma; 3. No positive lymph nodes in unilateral or bilateral regions III and IVa; 4. Clinical stage I-IVa (AJCC/UICC 8th edition), with no evidence of distant metastasis; 5. Normal thyroid function; 6. ECOG performance status of 0-1; 7. Treatment-naïve patients who have not received any prior antitumor therapy; 6. No contraindications to radiotherapy or chemotherapy; 9. Adequate organ function, meeting the following criteria: Hematologic criteria: WBC ≥ 4.0 × 10⁹/L, ANC ≥ 1.5 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 90 g/L (no transfusion, blood products, or hematopoietic growth factors used within the past 7 days); Biochemical criteria: ALT and AST < 1.5 × ULN, ALP < 2.5 × ULN, total bilirubin < ULN, BUN and creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).

10. Voluntarily agreed to participate in the study, signed the informed consent form, demonstrated good compliance, and agreed to follow-up.

Exclusion Criteria:

1. History of other malignant tumors (excluding basal cell carcinoma/squamous cell carcinoma of the skin or cervical carcinoma in situ);
2. History of radiotherapy (excluding radiotherapy outside the planned target area for conditions such as melanoma);
3. History of neck surgery;
4. Any severe comorbidities that may pose risks to the study or affect compliance, such as unstable heart disease requiring treatment, kidney disease, chronic hepatitis, poorly controlled diabetes (fasting blood glucose > 1.5 × ULN), or psychiatric disorders;
5. History of hyperthyroidism, hypothyroidism, or immune-related thyroid disorders;
6. Other family or social factors, as judged by the investigator, may force the study's early termination, compromise patient safety, or affect the collection of trial data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional Recurrence-free Survival | 3 years
  Regional Recurrence-Free Survival (RRFS) is defined as the time interval from the date of randomization to the date of lymph node failure in the cervical lymphatic drainage area or the last follow-up date.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Overall Survival (OS) is defined as the time interval from the date of randomization to the date of death from any cause or the last follow-up date.
Disease-free Survival | 3 years
  Disease-Free Survival (DFS) is defined as the time interval from the date of randomization to the date of tumor recurrence or death from any cause.
Hypothyroidism-Free Survival | 3 years
  Hypothyroidism-free survival is defined as the time interval from the date of randomization to the date of the first occurrence of hypothyroidism or the last follow-up date.
Clinical Hypothyroidism-Free Survival | 3 years
  Clinical hypothyroidism-free survival is defined as the time interval from the date of randomization to the date of the first occurrence of clinical hypothyroidism or the last follow-up date.
Global Health Status | 1year, 2 year and 3 years
  The quality of life of patients in the two groups will be assessed using the EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China